CLINICAL TRIAL: NCT01235481
Title: Validation of an Exercise DVD for Maintenance After 12-week Outpatient Pulmonary Rehabilitation Program: a Randomized Clinical Trial.
Brief Title: Validation of an Exercise DVD for Maintenance After Pulmonary Rehabilitation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Capital Health, Canada (Other)
Responsible Party: Principal Investigator, Paul Hernandez, Principle Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA-RS/2011-159
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Lung Diseases
Keywords: pulmonary rehabilitation; exercise therapy; chronic lung disease; self-efficacy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise DVD (Experimental): Exercise DVD to be used by participants 30-60 minutes, once daily to facilitate maintenance exercise training
  Interventions: Device: Exercise DVD; Behavioral: Usual Care
- Usual Care (Other): Participants advised to perform maintenance exercise training 30-60 minutes, once daily without benefit of exercise DVD
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Device: Exercise DVD — Exercise DVD added to usual care during maintenance phase of pulmonary rehabilitation
  Other Names: Home exercise training
  Arms: Exercise DVD
Behavioral: Usual Care — Usual care during maintenance phase post pulmonary rehabilitation
  Other Names: No exercise DVD provided

SUMMARY:
The Public Health Agency of Canada estimates that over 3.5 million Canadians live with chronic respiratory diseases, such as COPD (chronic bronchitis and emphysema), asthma, sleep apnea, and lung cancer. Nova Scotia has been reported to have one of the highest rates of chronic lung disease among Canadian provinces, likely a reflection of both the age of the population and high rates of exposures to occupational dusts and smoking. Pulmonary rehabilitation is a multidisciplinary intervention, involving exercise and education for patients with chronic lung disease. Pulmonary rehabilitation has been demonstrated to improve patient symptoms, exercise capacity, and quality of life while reducing health resource utilization. Many studies have shown that the benefits of pulmonary rehabilitation tend to diminish over time after program completion. The best interventions to maintain the benefits of pulmonary rehabilitation remain unclear.

The purpose of this study is to validate incorporation of an exercise DVD into a maintenance program after pulmonary rehabilitation. 100 subjects will be recruited over 2-years from pulmonary rehabilitation programs at Capital Health, with 50 individuals randomized to usual care following PR and 50 individuals randomized to usual care plus the exercise DVD. Study subjects will be evaluated at time of enrolment in pulmonary rehabilitation, at completion of pulmonary rehabilitation and 6-months post- pulmonary rehabilitation. Study outcome measures will include exercise capacity, exercise compliance, health-related quality of life, confidence with performing exercise, and satisfaction with the exercise DVD. The primary outcome measure will be a change in functional exercise capacity as determined by the distance walked in 6-minutes, a commonly used and validated assessment tool for patients with chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* any participant enrolled in pulmonary rehabilitation program

Exclusion Criteria:

* Patients who do not have access to a DVD player.
* Inability to commit to the study plan.
* Cognitive or language barriers interfering with completion of the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
6MWD | 6 months

SECONDARY OUTCOMES:
disease-specific quality of life (CRQ) | 6 months
exercise compliance | 6 months
exercise self-efficacy | 6 months
subject satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hernandez, MDCM, FRCPC, Principal Investigator — Queen Elizabeth II Health Sciences Centre
Locations (2):
- Canada (2):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cobequid Community Health Centre, Lower Sackville, Nova Scotia